CLINICAL TRIAL: NCT02904304
Title: National Clinical Trial,Phase III, Multicenter, Randomized, Prospective, Double-blind, Parallel, Placebo-controlled, to Evaluate the Efficacy, Safety and Superiority of Decongex Gripe in the Treatment of Symptoms Associated With Common Cold
Brief Title: Desloratadine,Phenylephrine Hcl,Ibuprofen Compared to Placebo in Treatment of Symptoms Associated With Common Cold/Flu
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: the viability of the study is being analyzed
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-DNT-03(02/16)
Record Dates: First submitted 2016-03-08; First posted 2016-09-16 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Cold
Keywords: Flu; Treatment
MeSH Terms: conditions — Common Cold; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desloratadine+Phenylephrine+Ibuprofen (Experimental): It's a tablet manufactured by Aché S.A., composed of desloratadine 2,5mg, Phenylephrine hydrochloride 20mg and Ibuprofen 400mg.
  Tablet will be dispensed in a cartridge containing 10 tablet to 75 participants.
  Interventions: Drug: Desloratadine+Phenylephrine+Ibuprofen
- Placebo (Placebo Comparator): It's a tablet manufactured by Aché S.A,. composed of placebo will be dispensed in a cartridge containing 10 tablet to 75 participants. The participants shall administer the placebo tablets to enable the double-blind study.
  The use of placebo comparator is important in this type of pathology because with this design will be able to evaluate the response of the pure treatment, rapid relief of symptoms, or 03 hours after the first administration of study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desloratadine+Phenylephrine+Ibuprofen — 01 tablet, orally, every 12 hours.
  Other Names: Desloratadine+Phenylephrine hydrochloride+Ibuprofen
  Arms: Desloratadine+Phenylephrine+Ibuprofen
Drug: Placebo — 01 tablet, orally, every 12 hours.
  Arms: Placebo

SUMMARY:
National clinical trial, phase III, multicenter, randomized, prospective, double-blind, parallel, placebo-controlled, which one hundred and fifty (150) subjects of both sexes aged equal or more than 18 years will be randomly allocated to one the drug group or placebo group.

DETAILED DESCRIPTION:
The investigational product is a combination of desloratadine, phenylephrine hydrochloride and ibuprofen.

The desloratadine is a antihistamine and selectively block the activity of histamine receptor-1 (H1) resulting in a non sedative and prolong antiallergic effect.

The phenylephrine is a potent stimulator of the postsynaptic α receptor with minimal effect on β receptors in the heart.

The ibuprofen's mechanism is not fully known. It is a non selective inhibitor of cyclooxygenase, an enzyme that is involved in prostaglandin synthesis by the route from arachidonic acid. It is believed that the pharmacological effects are due to inhibition of cyclooxygenase-2 (COX-2), which reduces prostaglandin synthesis involved in the mediation of inflammation, pain, fever and swelling.

ELIGIBILITY:
Inclusion Criteria:

* Age older or equal to 18 and younger than 66 years;
* Subjects diagnosed with common cold / flu syndrome defined by clinical evaluation and the presence of two or more of the following symptoms: sneezing, rhinorrhea, nasal obstruction, headache, throat discomfort, sore throat, dysphonia, myalgia, cough and fever classified as moderate or intense in four intensity scale (04) items (0 = absent, 01 = light, 02 = moderate, 03 = severe);
* Beginning of the symptoms of common cold / flu-like syndrome in a minimum period of 24 hours and a maximum of 72 hours prior to V0;
* Ability to understand and consent to participate in this clinical research, expressed by signing the Informed Consent Form (ICF);

Exclusion Criteria:

* Any laboratorial finding (clinical evaluation / physical evaluation / vital signs / ECG changes) that the Investigator consider a risk to subject of the study;
* Hypersensitivity to the drug components used during the study;
* Women in pregnancy or nursing period;
* Women in reproductive age who do not agree to use contraception acceptable [oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch and tubal ligation]; other than surgically sterile (bilateral oophorectomy or hysterectomy), postmenopausal for at least one (01) years or sexual abstinence;
* Subjects that has participated in clinical trial protocols in the last twelve (12) months (National Board of Health- Resolution 251 of 07 August 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
* Alcohol abuse that, according to the investigator, may interfere with the pharmacological adherence to the clinical protocol;
* Any medical conditions which may interfere with efficacy and / or safety of the treatment with the investigational product, such as but not limited to disorders described below:
* Untreated or uncontrolled Hyperthyroidism
* Uncontrolled epilepsy
* diagnosis of glaucoma
* Moderate or severe persistent asthma (untreated or uncontrolled)
* NSAID-induced asthma diagnosed
* Systemic hypertension (SH) stage III uncontrolled
* Moderate and severe congestive heart failure
* Acute myocardial infarction
* unstable angina
* Uncontrolled cardiac arrhythmia
* Liver failure with clinical consequences
* Renal failure with clinical consequences
* Diagnosed HIV positive
* uncontrolled Diabetes type 1 or type 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the superiority of Desloratadine + Phenylephrine + Ibuprofen over placebo | 03 hours after the first dose
  To evaluate the association of the superiority fixed dose of desloratadine 2.5mg, 20mg phenylephrine hydrochloride and ibuprofen 400 mg compared to placebo in the treatment of symptoms related to the common cold / flu syndrome by varying the intensity total score of symptoms, three (03 ) hours after the first dose of investigational product.

SECONDARY OUTCOMES:
Evaluation of the symptoms related to the common cold / flu syndrome. | 02 days after initiation of treatment, compared to baseline.
  Absolute variation in total score intensity of symptoms related to the common cold / flu-like symptoms 02 days after the start of treatment compared to baseline.
Satisfaction of the quality of sleep | On the first day and on the second day after the start of treatment.
  Distribution of subjects in each treatment group as their perception to the sleep quality, assessed at baseline by answering the following statement: " Last night, with this cold, I did not sleep as well as I usually sleep "based on a scale of 0 to 4 points (0 = strongly disagree, 1 = disagree, 2 = neither agree nor disagree, 3 = agree and 4 = I totally agree).
The need for use of the rescue medication measured through the subject's diary. | On the first day and on the second day after the start of treatment.
  Proportion of subject in each treatment group who used at least once the rescue medication (Tylenol®) in the first (Day 01) and on the second day (day 02) after treatment, measured through the subject's diary.
The need for use of the rescue medication according to accounting of rescue medication returned. | On the first day and on the second day after the start of treatment.
  Proportion of subject in each treatment group who used at least once the rescue medication (Tylenol®) in the first (Day 01) and on the second day (day 02) after treatment, accounting of rescue medication (Tylenol®) returned.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Crippa Jr., Principal Investigator — Allergisa Pesquisa Dermato-Cosmética Ltda
Locations (1):
- Allergisa Pesquisa Dermato Cosmética Ltda., Campinas, São Paulo, Brazil